CLINICAL TRIAL: NCT05172674
Title: Ultrasound Diagnosis of Placental and Umbilical Cord Anomalies in Singleton Pregnancies Resulting From In-vitro Fertilization: a Prospective Cohort Study
Brief Title: Ultrasound Diagnosis of Placental and Umbilical Cord Anomalies in Singleton Pregnancies Resulting From In-vitro Fertilization
Acronym: PLACENTA
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 20/2019/Oss/AOUBo
Record Dates: First submitted 2021-12-13; First posted 2021-12-29 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Placenta Diseases; IVF
MeSH Terms: conditions — Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spontaneous pregnancies
  Interventions: Diagnostic Test: ultrasound according routine antenatal care
- pregnancies arising through IVF (homologus + hetereologus)
  Interventions: Diagnostic Test: ultrasound according routine antenatal care

INTERVENTIONS:
Diagnostic Test: ultrasound according routine antenatal care — ultrasound examinations at 11-14, 19-22 and 33-35 weeks

SUMMARY:
Objectives: to identify which type of placental and umbilical cord abnormalities are more common in IVF singleton pregnancies; to investigate if heterologous fertilization is an additional risk factor for the development of these abnormalities.

Methods: this was a multicenter prospective cohort study study involving two tertiary centres (S. Orsola Hospital, University of Bologna and Institute for Women's Health, University College of London). Patients with a singleton pregnancy conceived with IVF were consecutively recruited between May 2019 to January 2021. Each case was matched with a control presenting with a spontaneous pregnancy during the same period of time. All patients underwent similar antenatal care, which included ultrasound examinations at 11-14, 19-22 and 33-35 weeks. Ultrasound findings of placental and/or umbilical cord abnormalities were recorded in the two groups and confirmed after birth. The incidence of placental/cord findings in the study group was assessed using the chi-squared test or Fisher's exact test, where appropriate. Post-hoc pairwise comparisons were performed with the Fisher's exact test, using the Simes' method for false discovery rate control.

DETAILED DESCRIPTION:
This was a multicenter prospective cohort study study involving two tertiary centres (S. Orsola Hospital, University of Bologna and Institute for Women's Health and University College of London). All patients with a singleton pregnancy conceived with IVF were consecutively recruited between 1st of May 2019 to 31st March 2021. Each case was matched with a control presenting with a SC during the same period of time.

All patients had antenatal care using a similar clinical protocol, which included at 11-14 weeks (nuchal thickness screening scan), 19-22 weeks (detailed fetal anatomy scan) and 33-35 weeks (growth scan). All ultrasound examinations are carried out transvaginally and/or transabdominally by experienced operators using a high-resolution ultrasound equipment. Ultrasound findings of placental and/or umbilical cord abnormalities were recorded in each case using a standardized reporting protocol including placental location, cord insertion. The placenta was recorded as "low lying" when the edge was 0.5-2 cm from the internal os of the uterine cervix. When the placenta was <0.5cm from the internal os or completely covering it, it was defined as placenta previa (marginal or complete). Ultrasound signs of PAS were recorded using the standardized description proposed by the EW-AIP including for grey scale imaging: loss of clear zone, myometrial thinning, the presence of placental lacunae; bladder wall interruption; placental bulge and focal exophytic mass and for CDI: utero-vesical hypervascularity; subplacental hypervascularity; bridging vessels and lacunae feeder vessels. Additional transabdominal and transvaginal sonographic (TVS) examinations of the placenta and cord insertion were performed at 28-30 weeks and 35-36 weeks when anomalies were identified at the 19-22 weeks scan.

Women with multiple pregnancies or requiring emergency delivery before 32 weeks were excluded from the study group. All patients were managed according to local protocols.

Patient's demographic data, previous obstetric and gynecological history, clinical findings, ultrasound data and images and symptoms at the time of the first examination were recorded and stored in a specialized database (Viewpoint Version 5, Bildverargeritung GmbH, Munich, Germany). All placentas were examined at delivery by the obstetric team and histopathological evaluation has been carried out when clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* spontaneous pregnancies or pregnancies conceived with IVF

Exclusion Criteria:

* multiple pregnancies

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients with a singleton pregnancy conceived with IVF were consecutively recruited between 1st of May 2019 to 31st March 2021. Each case was matched with a control presenting with a SC during the same period of time.
  All patients had antenatal care using a similar clinical protocol, which included at 11-14 weeks (nuchal thickness screening scan), 19-22 weeks (detailed fetal anatomy scan) and 33-35 weeks (growth scan).
Sampling Method: Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
type of placental and umbilical cord abnormalities | 8 months
  to identify which type of placental and umbilical cord abnormalities are more common in IVF singleton pregnancies
heterologous fertilization | 8 months
  to investigate if heterologous fertilization is an additional risk factor for the development of these abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
we could share all IPD that underlie results in a publication